CLINICAL TRIAL: NCT00459615
Title: A Phase II, Randomized, Open-Label, Dose-Ranging Study of Intravenous Artesunate Therapy for the Treatment of Acute, Uncomplicated Plasmodium Falciparum Malaria.
Brief Title: Phase II Dose Ranging Study of Artesunate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Office of the Surgeon General (U.S. Federal Agency)
Collaborators: Military Infectious Diseases Research Program (MIDRP) (Network); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Organization: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WRAIR 1263; HSRRB Protocol Log#A-13912a,b
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Falciparum Malaria; Uncomplicated Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; Injections

INTERVENTIONS:
Drug: Artesunate for Injection

SUMMARY:
The purpose of this study is to compare four regimens using US FDA GMP intravenous artesunate for the treatment of uncomplicated Plasmodium falciparum malaria to identify the most effective treatment regimen as determined by rapidity of parasite clearance by microscopy.

DETAILED DESCRIPTION:
To compare the efficacy and tolerability of intravenous artesunate for the initial treatment of uncomplicated Plasmodium falciparum malaria at doses that bracket anticipated clinical doses (2.4 mg/kg once daily for 3 days; or 2.4 mg/kg initially, at 12 hours on Day 0, and then daily on Day 1 and 2) and thereby establish the safest, highly efficacious dosing regimen for use in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic Plasmodium falciparum malaria infection as determined by malaria smear with a parasite density of ≥ 5000 asexual parasites/mL
2. Age: 5-65 year old males and females.
3. Written informed consent must be obtained from adults age > 18 years. Parental consent will be obtained from children and adolescents, and subject assent will also be obtained from adolescents (age 12-17 years).
4. Willing to stay hospitalized for 4 days for treatment and for 3 scheduled follow-up outpatient visits at Day 7, 14 and 28.

Exclusion Criteria:

1. Pregnant women (clinically or by positive urine β-HCG) and nursing mothers
2. Clinical evidence of severe malaria (see Appendix B)
3. Mixed malaria infection on admission by malaria smear
4. A previous history of intolerance or hypersensitivity to the study drug artesunate or other artemisinin derivatives or Malarone.
5. Efficacious malaria drug therapy administered in the past 30 days by history (i.e. quinine, mefloquine, lumefantrine and artemisinin derivatives)
6. Previous participation in this trial or participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study.
7. Laboratory evidence or a history of significant liver or renal functional abnormality.
8. Anyone who has received a transfusion or any blood product within 30 days
9. Unable and/or unlikely to comprehend and/or follow the protocol.
10. Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this pharmacodynamic study is clearance of falciparum parasites from the blood.
Reference microscopic interpretation of Giemsa-stained thick and thin blood smears for malaria will serve as the diagnostic method of parasitemia detection.
Parasite clearance will be quantified using a discrete variable denoting efficacy to clear at least 90% of asexual parasites from the peripheral blood by 48 hours after administration of IV artesunate

SECONDARY OUTCOMES:
Additional measures of parasite clearance will also be assessed.
A continuous variable of time to parasite reduction milestones:
parasite clearance time (PCT90 and PCT100), and parasite reduction ratios (PRR12h and PRR24h) at defined time points , and
A continuous variable of area under the curve (AUC) of quantifiable parasitemia
Tolerability of the treatment regimens will also be assessed throughout the study through use of evaluation for adverse events and safety laboratories to include hematology and chemistry tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polhemus, MD, Principal Investigator — USAMRU-K; Bryan Smith, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (2):
- New Nyanza Provincial Hospital, Kisumu, Nyanza, Kenya
- Kwai River Christian Hospital, Sangkhla Buri, Kanchanaburi, Thailand

REFERENCES:
- See also: Related Info — http://usamrukenya.org